CLINICAL TRIAL: NCT03234920
Title: Effects of Beta-hydroxy-beta-methylbutyrate (HMB) Supplementation After Liver Transplantation: Randomized and Controlled Pilot Study
Brief Title: Beta-Hydroxy-Beta-Methylbutyrate (HMB) Supplementation After Liver Transplantation
Acronym: HMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Manuela Merli, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URomLSHMB
Record Dates: First submitted 2017-07-17; First posted 2017-08-01 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Sarcopenia
Keywords: cirrhosis; liver transplantation; HMB
MeSH Terms: conditions — Sarcopenia; Fibrosis | interventions — beta-hydroxyisovaleric acid

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- Control Group (Placebo Comparator): Placebo The placebo will be 200 ml of fruit juice twice a day. Placebo will be provided for 12 weeks
  Interventions: Other: Placebo
- Group 2 - Treatment group (Experimental): HMB Supplementation with 1.5 g of HMB dissolved in 200 ml of fruit juice and taken twice daily. Supplementation will be provided for 12 weeks
  Interventions: Dietary Supplement: BETA-HYDROXY-BETA-METHYLBUTYRATE (HMB)

INTERVENTIONS:
Dietary Supplement: BETA-HYDROXY-BETA-METHYLBUTYRATE (HMB) — 1.5 g of HMB dissolved in 200 ml of fruit juice will be provided for 12 weeks twice daily
  Arms: Group 2 - Treatment group
Other: Placebo — The placebo will be 200 ml of fruit juice given twice daily
  Arms: Group 1- Control Group

SUMMARY:
Sarcopenia is an independent predictor of morbidity and mortality in cirrhotic patient before and after liver transplantation. Beta-hydroxy-beta-methyl butyrate (HMB) is a leucine metabolite with potential efficacy in increasing protein synthesis, muscle mass and its functionality.

The aim of this randomized controlled study is to evaluate the effect of a nutritional supplementation with HMB after liver transplantation both on muscle mass and on muscle function.

DETAILED DESCRIPTION:
Protocol

1. Introduction:

   Sarcopenia, a condition of skeletal muscle mass depletion and reduction of muscle strength, is the most important aspect of malnutrition secondary to liver cirrhosis. Sarcopenia is recognized to be an independent factor of morbidity and mortality befor and after liver transplantation. The prevalence of sarcopenia in liver transplanted patients has been reported to vary between 40% and 76%. Sarcopenia in hepatic cirrhosis occurs as a result of an increase in proteolysis or a reduction in protein synthesis, or a combination of the two mechanisms. The alterations in the molecular pathways that regulate these mechanisms are not entirely known. Recent studies reported an increased expression of myostatin, a member of the transforming growth factor ß superfamily , in skeletal muscles of animal models with liver cirrhosis and in plasma of cirrhotic patients. The authors suggested that the increased expression of myostatin resulted in protein synthesis inhibition. In addition, myostatin is able to activate AMPK protein kinase, a signaling inhibitor of mTOR (mammalian target of rapamycin), key regulator of protein synthesis.

   After Liver transplant, secondary to the recovery of liver function, the progressive increase in caloric intakes and the increase in daily physical activity, an improvement in the nutritional status of the patient and normalization of body composition is expected. However, available data on the modification of nutritional status after liver transplantation do not confirm the expected results: worsening of nutritional status was reported in the perioperative period with further depletion of lean mass as a result of surgical stress, bed rest and postoperative complications. A lack of recovery of muscle mass was documented even after one year of transplantation.

   Molecular mechanisms responsible for sarcopenia after liver transplantation are not fully clarified. The only study on a small sample of muscle biopsies in post-transplant patients described a persistent increase in myostatin expression in these patients. The immunosuppressive therapy used in the post transplant involves the use of calcineurin inhibitors, a protein involved in differentiation and hypertrophy of muscle fibers, mTOR inhibitors and corticosteroids. The use of these drugs is another factor contributing to sarcopenia after transplantation.

   o HMB: HMB is a metabolite of leucine with the potential to increase performance and muscle trophism. Studies in experimental models of cachexia have resulted in increased phosphorylation and activation of secondary mTOR after use of HMB. Experimental studies performed on myoblastic cell cultures also revealed an increased expression of IGF-1 secondary to HMB treatment. Such evidence confirms the anabolic properties of the HMB. HMB has also been shown to suppress proteolysis by inhibition of the ubiquitin-proteasome pathway in models of neoplastic cachexia and to eb effective in reducing muscular atrophy secondary to steroid therapy. The association of anti-proteolytic and anabolic properties targeting mTOR make HMB a potentially effective supplement for the treatment of sarcopenia after liver transplantation. There are currently no data on the use of HMB in this category of patients.
2. Aims of the study:

   Primary aim of the study: Evaluate the therapeutic efficacy of HMB supplementation for three months in patients undergoing liver transplantation on recovery of skeletal muscle mass shortly after transplantation (third to fourth month after transplantation).

   Secondary aims of the study:
   * Evaluate the therapeutic efficacy of HMB supplementation for three months in patients undergoing liver transplantation on recovery of skeletal muscular function shortly after transplantation (third to fourth month after transplantation).
   * Evaluate the long-term effects of HMB supplementation in terms of recovery of skeletal muscle mass (6 and 12 months after transplantation).
   * Evaluate the possible effect of HMB supplementation on post-transplant morbidity (hospitalization, infectious complications, onset of metabolic complications).
   * Evaluate tolerance for HMB intake in liver transplant patients

   This controlled trial is not sponsored by a drug company.
3. Patients:

   The protocol of the study needs to be approved by the local ethic committee. Patients are enrolled in the study after been informed of the purpose and protocol of treatment and need to sign a written informed consent.
4. Statistical analysis, sample size and randomization:

   For categorical variables, the Person-Chi-square test or the Fischer test will be used. For continuous variables, the Mann-Whitney Test will be used. The ANOVA variance analysis will be applied followed by the "t-test" when significant differences will be highlighted. Values of p <0.05 will be considered statistically significant.

   For the sample size calculation, the increase in muscle mass, evaluated by DEXA and expressed as Fat Free Mass Index-FFMI (core indexed for height), 12 weeks after the beginning of supplementation was considered as the primary endpoint. On the basis of literature data, the investigators expect unchanged lean mass in the control group with a DS of ± 1 kg / m2 at 3-4 months after supplementation. In the HMB-treated group the investigators expect to increase the FFMI of 1.2 kg / m2 with the same DS. A total of 12 patients per group will need to have a statistical power of at least 80% with an alpha error of 5%.Block randomization, consisting of 4 individuals per block, was executed in a 1:1ratio using random numbers generated by an independent statistician (SPSS version 16.0). Knowledge of the randomization code was limited to the physician.
5. Protocol of the study:

Basal Evaluation:

The registration will include the main clinical and biochemical data prior to transplantation (including nutritional evaluation if present) and after transplantation.

Nutritional counseling will be provided to all patients to ensure similar caloric and daily protein intake in the two groups, according to the current guidelines (caloric intake of 20-25 kcal / kg / die ± 10%, protein intake of 1.2 g / kg / day).

At the time of the enrollment and during the subsequent controls the following data will be recorded :

1. calorie intake in the week preceding the visit by a three days non-consecutive food diary;
2. anthropometric parameters (height, weight, body mass index, brachial circumference, triceps)
3. body composition by dual-energy-xray-absorptiometry (DEXA) using dedicated software to estimated fat free mass index (FFMI) (Fat free mass in kg/ height in cm)
4. muscular function evaluated by 6 minute walk test-6MWT, Timed Up and Go test-TUGT), e l'Hand grip Test (HG).
5. biochemical and metabolic parameters
6. pharmacological therapy

During the study, clinical complications (hospital admissions, infectious events, onset of comorbidity) will be recorded.

During the study, the tolerability of the supplement (analogue-visual scale), adherence to absorption and any intolerance or secondary adverse effects will be detected.

Randomization: Patient are randomized to Group 1 - placebo (or control group) and Group 2 - supplementation (or treatment group)

Randomization: Patient are randomized to Group 1 - placebo (or control group) and Group 2 - supplementation (or treatment group)

The placebo will be 200 ml of fruit juice given twice daily. Supplementation will be HMB 1.5 g dissolved in 200 ml of fruit juice and taken twice daily. Supplementation/placebo will be provided for 12 weeks.

End-points of the study:

* Recovery of FFMI ( 3°-4° after liver transplantation)
* Recovery of muscle function (amelioration of 6-MWT, TUGT test and HG test) (3-4°, 6° and 12th month after liver transplantation )
* Reduction of morbidity after liver transplantation (Hospital admission, infections, onset of metabolic disease) 3-4°, 6° and 12th month after liver transplantation )
* Tolerably of HMB supplementation ( 3°-4° after liver transplantation) Collateral effects of HMB are recorded.

ELIGIBILITY:
Inclusion Criteria:

* 1. Liver transplantation

Exclusion Criteria:

* 1. Multiple organ transplantation
* 2. Low compliance

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-09-25 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in Fat Free Mass Index 3-4 months after transplantation | 3-4° months after transplantation
  Increase of Fat Free Mass Index-FFMI (FFMI) evaluated by DEXA

SECONDARY OUTCOMES:
Changes in Fat Free Mass Index 6 and 12 months after transplantation | 6° and 12° months after transplantation
  Increase of Fat Free Mass Index-FFMI (FFMI) evaluated by DEXA
Changes in 6MWT at 3-4, 6 and 12 months after transplantation | 3°-4°, 6° and 12° months after transplantation
  Recovery of muscle mass function evaluated by minute walk test-6MWT
Changes in test-TUGT at 3-4, 6 and 12 months after transplantation | 3°-4°, 6° and 12° months after transplantation
  Recovery of muscle mass function evaluated by Timed Up and Go test-TUGT
Changes in HG Test at 3-4, 6 and 12 months after transplantation | 3°-4°, 6° and 12° months after transplantation
  Recovery of muscle mass function evaluated by Recovery of muscle mass function evaluated by Hand grip Test (HG)
Evaluation of days of hospitalization during the study period | 3°-4°, 6° and 12° months after transplantation
  Days of Hospitalization will be recorded
Evaluation of onset of metabolic syndrome after liver transplantation classified sec. APT III classification | 3°-4°, 6° and 12° months after transplantation
  onset of metabolic syndrome diagnosed by ATP III classification
Incidence of Treatment-Emergent Adverse Events evaluated to analog-visual scale | 3°-4°, 6° and 12° months after transplantation
  Tolerability of supplementation evaluated to analog-visual scale

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Merli, Prof, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Gastroenterology Department, Sapienza University of Rome, Rome, Italy

REFERENCES:
- [Background] Dasarathy S. Consilience in sarcopenia of cirrhosis. J Cachexia Sarcopenia Muscle. 2012 Dec;3(4):225-37. doi: 10.1007/s13539-012-0069-3. Epub 2012 May 31. PMID 22648736
- [Background] Merli M, Giusto M, Riggio O, et al. Improvement of nutritional status in malnourished cirrhotic patients one year after liver transplantation. eESPEN 2011 (2011) e1-e6
- [Background] Giusto M, Lattanzi B, Albanese C, Galtieri A, Farcomeni A, Giannelli V, Lucidi C, Di Martino M, Catalano C, Merli M. Sarcopenia in liver cirrhosis: the role of computed tomography scan for the assessment of muscle mass compared with dual-energy X-ray absorptiometry and anthropometry. Eur J Gastroenterol Hepatol. 2015 Mar;27(3):328-34. doi: 10.1097/MEG.0000000000000274. PMID 25569567
- [Background] Tsien C, Garber A, Narayanan A, Shah SN, Barnes D, Eghtesad B, Fung J, McCullough AJ, Dasarathy S. Post-liver transplantation sarcopenia in cirrhosis: a prospective evaluation. J Gastroenterol Hepatol. 2014 Jun;29(6):1250-7. doi: 10.1111/jgh.12524. PMID 24443785
- [Background] Aversa Z, Bonetto A, Costelli P, Minero VG, Penna F, Baccino FM, Lucia S, Rossi Fanelli F, Muscaritoli M. beta-hydroxy-beta-methylbutyrate (HMB) attenuates muscle and body weight loss in experimental cancer cachexia. Int J Oncol. 2011 Mar;38(3):713-20. doi: 10.3892/ijo.2010.885. Epub 2010 Dec 23. PMID 21184031
- [Background] Gerlinger-Romero F, Guimaraes-Ferreira L, Giannocco G, Nunes MT. Chronic supplementation of beta-hydroxy-beta methylbutyrate (HMbeta) increases the activity of the GH/IGF-I axis and induces hyperinsulinemia in rats. Growth Horm IGF Res. 2011 Apr;21(2):57-62. doi: 10.1016/j.ghir.2010.12.006. Epub 2011 Jan 14. PMID 21237681
- [Background] Aversa Z, Alamdari N, Castillero E, Muscaritoli M, Rossi Fanelli F, Hasselgren PO. beta-Hydroxy-beta-methylbutyrate (HMB) prevents dexamethasone-induced myotube atrophy. Biochem Biophys Res Commun. 2012 Jul 13;423(4):739-43. doi: 10.1016/j.bbrc.2012.06.029. Epub 2012 Jun 13. PMID 22705301